CLINICAL TRIAL: NCT05001919
Title: Concentrated Growth Factors Membrane in the Treatment of Intrabony Periodontal Defects in Localized Aggressive Periodontitis. A Randomized Controlled Split-Mouth Clinical Study
Brief Title: Concentrated Growth Factors in Treatment of Intrabony Defects in Localized Aggressive Periodontitis
Acronym: RCT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, malak mohamed shoukheba, associate prof, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Aggressive Periodontitis
Keywords: aggressive periodontitis; intrabony defect,; concentrated growth factors membrane
MeSH Terms: conditions — Aggressive Periodontitis

STUDY DESIGN:
Intervention Model Description: Twenty intra-bony defects in 10 patients were randomly assigned to either test or control group in split-mouth technique (10 sites in each group).
Who Masked: Participant, Outcomes Assessor
Masking Description: Investigator Malak. Shoukheba screened the patients and randomly assigned them to test and control groups and performed the treatment procedures for all participants. Investigator Ahmed. Bader recorded the clinical parameters and she was masked to the randomization for the extent of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- collagen membrane (Placebo Comparator): 10 sites treated with surgery and bone graft and collagen membrane as GTR
  Interventions: Procedure: GTR
- Concentrated growth factor membrane (Experimental): 10 sites treated by surgery +bone graft and concentrated growth factor membrane as GTR
  Interventions: Procedure: concentrated growth factor

INTERVENTIONS:
Procedure: GTR — intrabony defects treated by surgery and bone graft +collagen membrane
  Other Names: regenerative surgery
  Arms: collagen membrane
Procedure: concentrated growth factor — intrabony defects treated by surgery and bone graft +concenrated growth factor membrane
  Other Names: regenerative surgery
  Arms: Concentrated growth factor membrane

SUMMARY:
A total of 20 intra-bony defects in 10 LAP patients were randomly assigned into two groups 10 defects each in a split-mouth design. Group I treated by surgery plus Bio-Oss bone graft + collagen membrane (Control group). Group II, treated by surgery plus Bio-Oss bone graft + CGF membrane (Test group). Gingival index (GI), bleeding on probing (BOP), probing pocket depth and clinical attachment level (CAL) were assessed at baseline, 3, 6, and 12 months. Cone beam radiograph evaluation was taken at baseline, and 12 months after surgery..

DETAILED DESCRIPTION:
Full mouth scaling and root planing was done for all patients followed by Augmentin I gm and metronidazole 500 mg twice daily for 7 days. Additionally, Comprehensive oral hygiene instructions were given to the patients.

Sites grouping Four weeks following phase I therapy, the twenty defect sites were randomly classified by sealed envelopes into two groups ten each by a masked supervisor as follows: Group I (10 sites) received surgery + Bio-oss bone graft (Geistlich Pharma AG, Wolhusen, Switzerland) + collagen membrane (control group). Group II (10 sites) received surgery + Bio-oss bone graft +concentrated growth factors membrane (tested group).

After the administration of local anesthesia (Xylocaine 2% Adrenaline 1:80,000, ICPA, India), buccal and lingual sulcular incisions were made, and mucoperiosteal flaps were elevated. Thorough debridement of the defects was achieved with hand instruments. The surgical area was irrigated with copious amounts of sterile saline. Bio-oss granules were placed into the defects and the CGFs membrane was trimmed and adapted over the entire defect to cover 2-3 mm of the surrounding alveolar bone and to ensure the stability of the wound and the graft material. For control sites, Bio-oss grafts and a bioresorbable collagen membrane were trimmed and adjusted over the defect in such a way that the whole defect and 2-3 mm of the surrounding alveolar bone were completely covered. Then the flap was repositioned to achieve complete interproximal closure. The flap was then sutured with 4-0 absorbable sutures with single interrupted sutures. A periodontal pack was applied over the surgical area for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Presence of angular periodontal intra-bony defects with clinical attachment loss ≥5 mm measured from CEJ to the deepest propping depth with no evidence of gingival recession
* optimal compliance as evidenced by no missed treatment appointment and high attitude towards oral hygiene

Exclusion Criteria:

* Patients with relevant medical conditions that may affect periodontal regeneration and surgery
* smokers, pregnant or lactating women
* those whom periodontal surgery had previously been carried out on the selected site,
* and patients who taking any drug known to affect the number or function of platelets

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
probing pocket depth | 12 months
  measured from the gingival margin to the base of the pocket using periodontal probe in mm
clinical attachment level | 12months
  measured from the cemento-enamel junction to the base of the pocket using periodontal probe in mm
radiographic defect area by cone beam x ray | 12 months
  measured in square millimeter from cone beam x ray
radiographic bone density by cone beam | 12 months
  By Hounsfield unit from the cone beam x ray

SECONDARY OUTCOMES:
bleeding on probing | 12 months
  bleeding on probing according to Ainamo and Bay1975
gingival index | 12 months
  gingival index measured according to Loe and Silness 1963

CONTACTS AND LOCATIONS:
Locations (1):
- Malak Yousef Mohamed Shoukheba, Tanta, Egypt